CLINICAL TRIAL: NCT06056908
Title: Shwachman Diamond Syndrome Registry and Study (SDS Registry)
Brief Title: Shwachman Diamond Syndrome Registry and Study
Acronym: SDSR
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Akiko Shimamura, Director, Bone Marrow Failure and Myelodysplastic Syndrome Program, Boston Children's Hospital
Other Study IDs: P00020466
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Shwachman-Diamond Syndrome; Shwachman-Diamond Syndrome-Like
Keywords: Bone marrow failure; Inherited bone marrow failure syndromes; Bone marrow; Neutropenia; Leukemia; MDS; Pancreas; Cancer predisposition
MeSH Terms: conditions — Shwachman-Diamond Syndrome; Bone Marrow Failure Disorders; Congenital Bone Marrow Failure Syndromes; Neutropenia; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Years
Biospecimen Retention: Samples With DNA — Peripheral blood, bone marrow, skin cells, saliva or a buccal swab, and discards from clinical procedures may be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with SDS/SDS-Like conditions and their families

SUMMARY:
Shwachman-Diamond syndrome (SDS) is a genetic condition characterized by bone marrow failure, medical co-morbidities, and leukemia predisposition. SDS-Like patients share clinical features with SDS but lack mutations in known SDS genes. Since SDS/SDS-Like syndromes are rare diseases, data are sparse regarding the clinical features, natural history, clinical outcomes with current management, and treatment. For this reason, the SDS Registry was formed to collect clinical data from medical records and to bank biological samples with the goal of understanding SDS/SDS-Like diseases to develop better treatments and improve the health of patients with these conditions.

DETAILED DESCRIPTION:
The Shwachman-Diamond Syndrome Registry (SDSR) is dedicated to accelerating research and treatment for SDS to improve survival and quality of life for all patients with the disease. The SDSR is run jointly by Boston Children's Hospital and Cincinnati Children's Hospital Medical Center.

Objective and Aims:

The long term goals of the Registry are to improve diagnosis, inform medical management, and to develop better treatments for SDS and SDS-Like disorders.

To achieve these objectives, the Registry has the following specific aims:

* Characterize the natural history, medical complications, and treatment outcomes for patients with SDS and SDS-Like disorders.
* Investigate the molecular and genetic pathogenesis of SDS/SDS-Like conditions and their complications such as marrow failure and clonal evolution.
* Identify new genes causing SDS/SDS-Like conditions.
* Provide education on the diagnosis, medical management and treatment of SDS for patients, families and the medical/scientific community.

Methods: The SDSR collects information from medical records and biological samples. Samples for the SDSR are collected when they are obtained for clinical care so that no extra visits or procedures are needed. These samples may include blood, bone marrow, skin cells, saliva, or discards from other clinical procedures. Family members may also contribute blood samples. All information obtained by the SDSR is housed on a secure, HIPAA-compliant database. No personal information is shared outside of the study team.

ELIGIBILITY:
Inclusion Criteria: Shwachman Diamond syndrome, Shwachman-Diamond Syndrome-Like conditions, or a genetically undefined condition that shares clinical features with Shwachman Diamond Syndrome.

* Biallelic mutations in SBDS, or pathogenic mutations in DNAJC21, EFL1, or SRP54 OR
* Shwachman-Diamond Syndrome defined clinically OR
* Clinically suspected Shwachman-Diamond Syndrome OR
* Phenotypic features suggestive of SDS OR
* Parents, siblings, and other blood relatives of any age, living and deceased, of patients with SDS or SDS-Like conditions are eligible for this study

Exclusion Criteria:

• Patients with other diagnosed causes of bone marrow failure, exocrine pancreatic insufficiency and cancer predisposition will be excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known or suspected SDS or SDS-Like conditions and their relatives are eligible for the study. Patients may indicate interest in participation by contacting the registry team through the website at www.sdsregistry.org.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-01-19 (Actual); Primary Completion 2090-01-01 (Estimated); Study Completion 2090-01-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the natural history, medical complications, and treatment outcomes for patients with SDS and SDS-Like conditions. | 50 years
  The SDSR will collect clinical information regarding SDS and SDS-Like conditions. The goal is to understand the natural history, treatment outcomes and complications of these rare disorders in order to improve diagnosis, medical management, and treatment.
Investigate the molecular and genetic pathogenesis of SDS/SDS-Like condtions and their complications such as marrow failure and clonal evolution. | 50 years
  The SDSR will coordinate a repository of blood, cord blood, bone marrow, saliva, skin fibroblast, and tumor samples and cell lines from patients with SDS and SDS-Like conditions for basic science studies of molecular and genetic pathways causing these disorders and their complications. We will also study how genetic/molecular pathways may be targeted or corrected for the development of new therapies. To this end, we will create immortalized cell lines including EBV-transformed lymphoblasts, immortalized fibroblasts, and induced pluripotent stem cells. These cell lines will provide a renewable source of rare patient-derived material for these studies.
Identify new genes causing SDS/SDS-Like conditions | 50 years
  The SDSR will sequence DNA from patient samples to try to identify new genes that are involved in SDS/SDS-like phenotypes.
Provide education on the diagnosis, medical management, and treatment of SDS/SDS-Like conditions for patients, families, and the medical/scientific community. | 50 years
  The SDSR will disseminate information through the study website, conferences, and other scientific publications.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for the SDS Registry — https://www.sdsregistry.org/